CLINICAL TRIAL: NCT02673866
Title: A Randomized Double-Blind Placebo and Active Controlled Parallel Group Study to Evaluate the Efficacy and Safety of DS-1971a for the Treatment of Diabetic Peripheral Neuropathic Pain (DPNP)
Brief Title: Study to Evaluate the Efficacy and Safety of DS-1971a for the Treatment of Diabetic Peripheral Neuropathic Pain (DPNP)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: reassessment of phase 2 study indication
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS1971-A-U202
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Neuropathic Pain; Diabetes
Keywords: Diabetic Peripheral Neuropathic Pain (DPNP); Diabetes; Pregabalin; Spontaneous Pain; Hyperalgesia; Allodynia; Average Daily Pain Score (ADPS); Pain Associated Sleep Interference
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus; Hyperalgesia | interventions — DS-1971a; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- DS-1971a 400 mg TID (Experimental): DS-1971a 400 mg three times per day (TID)
  Interventions: Drug: DS-1971a; Drug: placebo
- DS1971a 400 mg BID (Experimental): DS1971a 400 mg twice per day (BID)
  Interventions: Drug: DS-1971a; Drug: placebo
- DS1971a 100 mg BID (Experimental): DS1971a 100 mg BID
  Interventions: Drug: DS-1971a; Drug: placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- Pregabalin (Active Comparator): Pregabalin
  Interventions: Drug: placebo; Drug: pregabalin

INTERVENTIONS:
Drug: DS-1971a
  Arms: DS-1971a 400 mg TID; DS1971a 100 mg BID; DS1971a 400 mg BID
Drug: placebo
Drug: pregabalin — pregabalin
  Arms: Pregabalin

SUMMARY:
The hypothesis of this Phase 2 study is that at least 1 dose regimen of DS-1971a will demonstrate clinical superiority to placebo in managing pain associated with DPNP, and will be generally well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Body mass index (BMI) ≤ 40 kg/m2 at screening.
* Able to give written informed consent.
* Type 1 or 2 diabetes.
* HbA1c ≥ 7.0% and < 9% at screening.
* On a stable anti-diabetic medication regimen (unchanged dose over the last 3 months for diabetes) prior to screening (insulin therapy is acceptable); no recent (i.e., within the previous 6 months) hospitalizations due to noncompliance or uncontrolled diabetes or introduction of new medications.
* ADPS of ≥ 4 on the 11-point numeric rating scale (NRS) over the past 7 days prior to randomization (based on completion of at least 4 daily pain diaries during the 7-day baseline period prior to randomization).
* Painful distal symmetrical sensorimotor polyneuropathy diagnosed for at least 6 months (positive Douleur Neuropathique 4 [DN4] questionnaire at screening).
* Women of child bearing potential (WOCBP) must be willing to use double-barrier contraception for the entire study.
* Subjects who, in the judgement of the Investigator, are likely to be compliant during the study.

Exclusion Criteria:

* Clinically significant unstable neurologic, psychiatric, ophthalmologic, hepatobiliary, respiratory, or hematologic illness or unstable cardiovascular disease (e.g., severe hypotension, uncontrolled cardiac arrhythmia, or myocardial infarction) or any other concurrent disease within 12 months prior to screening that in the opinion of the Investigator would interfere with study participation or assessment of safety and tolerability.
* Subjects who present with active cancer or human immunodeficiency virus (HIV) infection.
* Creatinine clearance rate < 60 mL/min.
* Current diagnosis of epilepsy or any seizure disorder requiring chronic therapy with anti-epileptics.
* Diagnosis of mononeuropathy.
* Subjects who are at risk of suicide as defined by their responses to the C-SSRS or in the opinion of the Investigator. Note: Subjects answering "yes" to any of the questions about suicidal ideation/intent/behaviors occurring within the past 12 months must be excluded (C-SSRS Suicide Ideation section-Questions 1, 2, 3, 4, or 5; C-SSRS Suicidal Behavior section, any of the suicide behaviors questions). Such subjects should be referred immediately to a mental health professional for appropriate evaluation.
* Any major uncontrolled psychiatric disorders such as bipolar disorder, schizophrenia, or major depression.
* Abnormal liver function (aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 2.5 × upper limit of normal (ULN), bilirubin > 1.5 ULN).
* Subjects with history of gout, and/or urate nephrolithiasis, and/or with abnormally low serum uric acid (below the lowest laboratory reference range both in men and women) at baseline.
* Other sources of pain that may confound assessment or self-evaluation of DPNP such as disseminated osteoarthritis or rheumatoid arthritis.
* Neurologic disorders unrelated to diabetic peripheral neuropathy that may confound the assessment of DPNP.
* Amputation of lower extremity (including above- and below-knee amputation) due to diabetes mellitus.
* Unable or unwilling to discontinue current medications for chronic pain for the duration of the trial.
* Use of concomitant medications (i.e., opioids, tricyclic anti-depressives, and/or gamma retinoids) that may confound assessments of efficacy and/or safety.
* Inability or unwillingness to discontinue any other prohibited concomitant medications (see Section 5.6).
* Abuse or dependence on prescription medications, street drugs, or alcohol within the last year.
* Women who are pregnant or breast-feeding or intend to become pregnant during the study period.
* Known hypersensitivity to pregabalin or DS-1971a and/or known treatment failure on pregabalin.
* Subjects who are a family member of the Investigator or any associate, colleague, and employee assisting in the conduct of the study (secretary, nurse, technician).
* Subjects who cannot be contacted by phone in an emergency.
* Participated in another clinical study within 30 days prior to screening or is receiving other investigational agents.
* Subjects who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change in weekly Average Daily Pain Score (ADPS) | week 0 (Baseline) to Week 7

SECONDARY OUTCOMES:
Response rate, proportion of subjects with ≥ 30% or ≥ 50% reduction | week 0 (Baseline) to Week 7
  Response rate, defined as the proportion of subjects with ≥ 30% or ≥ 50% reduction
Effect of DS-1971a on Patient Global Impression of Change (PGIC) in neuropathic pain | week 7
  Effect of DS-1971a on Patient Global Impression of Change (PGIC) in neuropathic pain
Effect of DS-1971a on pain intensity and severity | week 7
  Effect of DS-1971a on pain intensity and severity as assessed by the Short-Form McGill Pain Questionnaire (SF-MPQ)
Effect of DS-1971a on pain intensity and severity | week 7
  Effect of DS-1971a on pain interference with daily activities as assessed by a modified Brief Pain Inventory Short Form (BPI-SF)
Change in Hospital Anxiety and Depression Scale (HADS) | week 0 (Baseline) to Week 7
  Change as assessed by the Hospital Anxiety and Depression Scale (HADS)
Change in pain-associated sleep interference score (ADSIS) | week 0 (Baseline) to Week 7
  Change in pain-associated sleep interference as assessed by average daily sleep interference score (ADSIS)
Changes in subject general health status | week 0 (Baseline) to Week 7
  Changes in subject general health status as assessed by the Short Form 36 (SF-36) questionnaire
number and severity of Adverse Events (AEs), clinical laboratory abnormalities, physical examinations, ECGs, vital signs | week 0 (Baseline) to Week 7
  number and severity of AEs, clinical laboratory abnormalities, physical examinations, 12-lead electrocardiograms (ECGs), and vital signs
change in Columbia-Suicide Severity Rating Scale (C SSRS) | week 0 (Baseline) to Week 7
  change in Columbia-Suicide Severity Rating Scale (C SSRS)
Effects of treatments on neuropathic pain components | week 7
  Effects of treatments on neuropathic pain components assessed with the Neuropathic Pain Symptom Inventory (NPSI)
change in weekly ADPS responder rate | week 7
  Effects of DS-1971a versus pregabalin (titrated to 300 mg daily) in weekly ADPS responder rate at Week 7
Rescue medication usage | week 0 through week 7
  Rate of rescue medication usage